CLINICAL TRIAL: NCT03768492
Title: A Phase 1, Randomized, Double Blinded, Placebo Controlled Study of the Safety and Efficacy of a Caffeine-based Antifibrosis Cream in Patients With Breast Cancer Undergoing Radiation Therapy
Brief Title: Study of the Safety and Efficacy of a Caffeine-based Antifibrosis Cream in Patients With Breast Cancer Undergoing Radiation Therapy
Acronym: ReDCoAT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-00309
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Carcinoma Breast
Keywords: Masectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine Based Cream (Experimental): caffeine based cream during and for 4 weeks following radiation
  Interventions: Drug: Caffeine anhydrous 5% added to Lipoderm Cream Base.
- Placebo (Placebo Comparator): placebo cream during and for 4 weeks following radiation
  Interventions: Other: Lipoderm Cream Base

INTERVENTIONS:
Drug: Caffeine anhydrous 5% added to Lipoderm Cream Base. — Caffeine USP Anhydrous 5 gm Ethoxy Digylco Reagent 10 ml Professional Compounding Centers of America (PCCA) Lipoderm Base 85 gm
  Arms: Caffeine Based Cream
Other: Lipoderm Cream Base — Professional Compounding Centers of America (PCCA) Lipoderm Base 85 gm
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether a caffeine-based cream can reduce the rates of reconstructive complications in patients with tissue expander based reconstruction requiring post-mastectomy radiation therapy when compared to a placebo cream.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically-confirmed carcinoma of breast (all subtypes are permitted)
* Patient has undergone mastectomy with tissue expander-based reconstruction and require post-mastectomy radiation therapy (PMRT) per the - Stage DCIS (0) -III breast cancer, excluding any patients with inflammatory breast cancer at presentation.
* Patient will receive irradiation of the chest wall. Additional fields to treat the regional nodes including the supraclavicular / axillary and/or internal mammary chains is allowed but not required. If a patient requires a boost field to the chest wall, scar and/or nodal region this is allowed.

Exclusion Criteria:

* Patient with skin changes or inflammatory carcinoma at presentation Patient has (cT4b-d)
* unhealed wound in the radiation field
* Patient has allergy to Caffeine
* Patient has systemic lupus erythematosus or scleroderma that increases the risk of radiation dermatitis development
* Patient will receive concurrent chemotherapy with radiation. (Patient is allowed to take concurrent hormonal therapy or Trastuzumab)
* Planned accelerated or hypofractionated fractionation.
* Previous radiation to the ipsilateral breast or chest wall or thoracic region.
* Anyone who will require bolus use during radiation (per physician discretion) as this will increase rates of acute toxicity interfering with measurement of the primary study endpoint.
* All pre-menopausal women will require a urine qualitative pregnancy test to exclude pregnancy. Pregnant women will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Standard Toxicity Scoring | 4 Years
  The US National Cancer Institute developed the Common Terminology Criteria for Adverse Events (CTCAE), which was formerly called the Common Toxicity Criteria (CTC), which is a standardized classification of adverse effects in cancer therapy. The current version 5.0 was released in 2017. The criteria uses a grading system of 1 to 5 (e.g. Grade 1 = mild and Grade 5 = death related to AE).

CONTACTS AND LOCATIONS:
Overall Officials: Naamit Kurshan Gerber, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Single-institution investigator initiated trial. We are not going to make our data available to others.